CLINICAL TRIAL: NCT02913105
Title: A Randomized, Patient and Investigator Blinded, Placebo Controlled, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of LMB763 in Patients With Non-alcoholic Steatohepatitis (NASH)
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of LMB763 in Patients With NASH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLMB763X2201
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-01

CONDITIONS: Non-alcoholic Steatohepatitis NASH
Keywords: Non-alcoholic Steatohepatitis; NASH; Fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LMB763 (Experimental): Oral dose once daily for 12 weeks (84 days)
  Interventions: Drug: LMB763
- Placebo (Placebo Comparator): Oral dose once daily for 12 weeks (84 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LMB763 — Hard Gelatin Capsules
  Arms: LMB763
Drug: Placebo — Hard Gelatin Capsule
  Arms: Placebo

SUMMARY:
The purpose of the present study is to assess the effects of LMB763 with respect to safety, tolerability, and on markers of liver inflammation in patients with NASH

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients, 18 years or older
* Written informed consent
* Presence of NASH by histologic evidence (liver biopsy) and elevated alanine aminotransferase (ALT), OR phenotypic diagnosis of NASH based on elevated ALT, BMI and diagnosis of Type 2 diabetes mellitus

Exclusion Criteria:

* Current use of obeticholic acid (OCA)
* New initiation GLP-1 agonists such as liraglutide, exenatide , lixisenatide, albiglutide or dulaglutide within 3 months of screening
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 5 days after stopping study medication
* Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening
* Clinical evidence of hepatic decompensation or severe liver impairment
* Previous diagnosis of other forms of chronic liver disease
* Uncontrolled diabetes mellitus
* History or current diagnosis of ECG abnormalities
* Patients with contraindications to MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (13):
  - Novartis Investigative Site, Culver City, California
  - Novartis Investigative Site, Cypress, California
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami Springs, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Newport News, Virginia
- Australia (2):
  - Novartis Investigative Site, New Lambton, New South Wales
  - Novartis Investigative Site, Nedlands, Western Australia
- Novartis Investigative Site, Tbilisi, Georgia
- Novartis Investigative Site, Amman, Jordan
- New Zealand (5):
  - Novartis Investigative Site, Papatoetoe, Auckland
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Tauranga
  - Novartis Investigative Site, Wellington
- Novartis Investigative Site, San Juan, Puerto Rico
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lugano
- United Kingdom (3):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 25 centers across 6 countries.
Pre-assignment Details: A total of 121 participants were enrolled in the study, and included in the safety population. Placebo data have been pooled from placebo treated participants from both cohorts (100 mg and 50 mg matching placebo).
Groups:
- LMB763 100 mg: LMB763 100 mg capsules, orally, once daily for 12 weeks (84 days) under fasted conditions (no food or drink for at least 6 hours).
- LMB763 50 mg: LMB763 50 mg (2 x 25 mg) capsules, orally, once daily for 12 weeks (84 days) under fasted conditions (no food or drink for at least 6 hours).
- Pooled Placebo: LMB763 100 mg or 50 mg matching placebo capsules, orally, once daily for 12 weeks (84 days) under fasted conditions (no food or drink for at least 6 hours).
Period: Overall Study
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Started | 37 | 44 | 40
Completed | 22 | 39 | 33
Not Completed | 15 | 5 | 7
Not completed — Adverse Event | 11 | 0 | 4
Not completed — Non-Compliance With Study Drug | 0 | 0 | 1
Not completed — Reason Not Specified | 3 | 1 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants that received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo | Total
Number analyzed (Participants) | 37 | 44 | 40 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (15.55) | 49.5 (8.45) | 51.6 (11.65) | 50.8 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 24 | 69
  Male | 15 | 21 | 16 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 10 | 30
  Not Hispanic or Latino | 27 | 33 | 28 | 88
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 3 | 4 | 9
  Black Or African American | 1 | 2 | 0 | 3
  Multiple | 1 | 1 | 3 | 5
  Native Hawaiian Or Other Pacific Islander | 1 | 0 | 1 | 2
  White | 32 | 37 | 31 | 100
  Other | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation as per Medical or scientific judgment. No statistical analysis was planned for this primary outcome measure.
Time Frame: From date of First Participant First Treatment until Last Patient Last Visit (up to Day 112 (End of Study (EOS))
Population: Safety analysis set included all participants that received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
Participants
  AEs | 35 | 37 | 33
  SAEs | 2 | 3 | 0

2. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) Levels
Description: ALT level assessment is one of the diagnostic parameters in Liver function test (LFT). Baseline was defined as the mean of ALT levels at baseline and pre-dose visits. Geometric Mean and Geometric Coefficient of Variation for change are based on log-transformed ratio to baseline (i.e., change from baseline in the log domain).
Time Frame: Baseline to Day 84 (Week 12)
Population: Pharmacodynamic (PD) analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. Number analyzed included participants with a value at both Baseline and that time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: units per liter (U/L)
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
units per liter (U/L)
  Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 40 | 33
  Baseline for Day 84 Analysis | 67.215 (30.8) | 48.114 (42.2) | 59.544 (39.5)
  Change from Baseline at Day 84: number analyzed (Participants) | 24 | 40 | 33
  Change from Baseline at Day 84 | 0.667 (33.8) | 0.702 (41.1) | 0.901 (25.5)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Test type: Other — Log transformed ratio to baseline was analyzed using a repeated measures model which included effects for treatment, visit, treatment by visit interaction, stratification factor (Body Mass Index (BMI) group), log-transformed baseline and log-transformed baseline by visit interaction. BMI was separated into two groups low BMI (Asian<30 and Non-Asian<35) and high BMI (Asian >=30 and Non-Asian>=35); p = 0.7489, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.97, 90% CI 2-sided [0.83 to 1.13]
Statistical Analysis 2: Comparison: LMB763 100 mg vs Pooled Placebo; Test type: Superiority — Log transformed ratio to baseline was analyzed using a repeated measures model which included effects for treatment, visit, treatment by visit interaction, stratification factor (BMI group), log-transformed baseline and log-transformed baseline by visit interaction. BMI was separated into two groups low BMI (Asian<30 and Non-Asian<35) and high BMI (Asian >=30 and Non-Asian>=35); p = 0.0005, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.72, 90% CI 2-sided [0.62 to 0.84]
Statistical Analysis 3: Comparison: LMB763 50 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0005, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.74, 90% CI 2-sided [0.65 to 0.85]

3. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) of LMB763
Description: No statistical analysis was planned for this outcome measure.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Days 1 and 42
Population: Pharmacokinetic (PK) analysis set included all participants with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug and with no protocol deviations that impact on PK data. Number analyzed is the number of participants with data available for analysis at specified time-point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LMB763 100 mg | LMB763 50 mg
Number analyzed (Participants) | 37 | 43
nanograms per milliliter (ng/mL)
  Day 1 | 3080 (1360) | 1290 (620)
  Day 42: number analyzed (Participants) | 23 | 42
  Day 42 | 2230 (1190) | 1290 (690)

4. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of LMB763
Description: No statistical analysis was planned for this outcome measure.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Days 1 and 42
Population: PK analysis set included all participants with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug and with no protocol deviations that impact on PK data. Number analyzed is the number of participants with data available for analysis at specified time-point.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | LMB763 100 mg | LMB763 50 mg
Number analyzed (Participants) | 37 | 43
hour (h)
  Day 1 | 2.00 [1.00 to 6.00] | 2.00 [1.00 to 6.08]
  Day 42: number analyzed (Participants) | 24 | 42
  Day 42 | 2.03 [1.00 to 6.03] | 2.02 [1.00 to 6.00]

5. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of LMB763
Description: No statistical analysis was planned for this outcome measure.
Time Frame: 0 to 96 hours post-dose on Days 1 and 42
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LMB763 100 mg | LMB763 50 mg
Number analyzed (Participants) | 37 | 43
h*ng/mL
  Day 1: number analyzed (Participants) | 37 | 42
  Day 1 | 11200 (4740) | 4360 (2350)
  Day 42: number analyzed (Participants) | 23 | 42
  Day 42 | 8570 (4120) | 5180 (2870)

6. Secondary Outcome: Accumulation Ratio (Racc) of LMB763
Description: The drug accumulation ratio (Racc) is the ratio of accumulation of drug going from a single dose to steady state with repeated administration.
  No statistical analysis was planned for this outcome measure.
Time Frame: Day 42
Population: PK analysis set included all participants with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug and with no protocol deviations that impact on PK data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | LMB763 100 mg | LMB763 50 mg
Number analyzed (Participants) | 24 | 42
ratio | 0.903 (0.472) | 1.31 (0.641)

7. Secondary Outcome: Change From Baseline in Percentage of Liver Fat as Measured by Magnetic Resonance Imaging (MRI)
Description: Participants were to undergo MRI twice (Baseline and End of Treatment) during the course of the study to quantitate liver fat. Baseline was defined as the last available measurement prior to the first dose. Geometric Mean and Geometric Coefficient of Variation for change are based on log-transformed ratio to baseline (i.e., change from baseline in the log domain).
Time Frame: Baseline to Day 84 (Week 12)
Population: PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. Number analyzed included participants with a value at both Baseline and that time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of liver fat
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 35 | 44 | 39
percentage of liver fat
  Baseline for Day 84 Analysis: number analyzed (Participants) | 22 | 41 | 32
  Baseline for Day 84 Analysis | 18.751 (37.4) | 17.715 (42.6) | 17.476 (73.9)
  Change from Baseline at Day 84: number analyzed (Participants) | 22 | 41 | 32
  Change from Baseline at Day 84 | 0.648 (29.3) | 0.681 (38.6) | 0.962 (22.2)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Test type: Other — Log transformed ratio to baseline was analyzed using an ANCOVA model which included effects for treatment, log-transformed baseline and stratification factor (BMI group). BMI was separated into two groups, low BMI (Asian<30 and Non-Asian<35) and high BMI (Asian =30 and Non-Asian=35); p = 0.5354, ANCOVA; Geometric Mean Ratios = 0.95, 90% CI 2-sided [0.83 to 1.09]
Statistical Analysis 2: Comparison: LMB763 100 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < .0001, ANCOVA; Geometric Mean Ratios = 0.68, 90% CI 2-sided [0.59 to 0.78]
Statistical Analysis 3: Comparison: LMB763 50 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < .0001, ANCOVA; Geometric Mean Ratios = 0.71, 90% CI 2-sided [0.63 to 0.80]

8. Secondary Outcome: Change From Baseline in Weight
Description: Baseline was defined as the last available measurement prior to the first dose.
Time Frame: Baseline to Days 28, 42, 56, 84 and 112 (EOS)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
kilogram (kg)
  Baseline for Day 28 Analysis: number analyzed (Participants) | 30 | 43 | 37
  Baseline for Day 28 Analysis | 99.07 (22.560) | 97.82 (17.829) | 95.47 (22.921)
  Change from Baseline at Day 28: number analyzed (Participants) | 30 | 43 | 37
  Change from Baseline at Day 28 | -0.78 (1.591) | -0.71 (1.725) | -0.17 (1.516)
  Baseline for Day 42 Analysis: number analyzed (Participants) | 27 | 43 | 34
  Baseline for Day 42 Analysis | 96.89 (22.135) | 97.82 (17.829) | 95.30 (23.465)
  Change from Baseline at Day 42: number analyzed (Participants) | 27 | 43 | 34
  Change from Baseline at Day 42 | -1.04 (1.683) | -1.08 (2.335) | -0.24 (1.677)
  Baseline for Day 56 Analysis: number analyzed (Participants) | 26 | 42 | 35
  Baseline for Day 56 Analysis | 97.07 (22.555) | 97.86 (18.043) | 95.71 (23.244)
  Change from Baseline at Day 56: number analyzed (Participants) | 26 | 42 | 35
  Change from Baseline at Day 56 | -1.39 (1.970) | -1.39 (2.188) | -0.26 (1.777)
  Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 40 | 34
  Baseline for Day 84 Analysis | 97.34 (23.370) | 97.11 (17.905) | 95.91 (23.563)
  Change from Baseline at Day 84: number analyzed (Participants) | 24 | 40 | 34
  Change from Baseline at Day 84 | -1.47 (2.169) | -2.02 (3.451) | -0.21 (1.989)
  Baseline for Day 112 (EOS) Analysis: number analyzed (Participants) | 22 | 39 | 33
  Baseline for Day 112 (EOS) Analysis | 98.74 (23.941) | 95.38 (14.810) | 95.85 (23.926)
  Change from Baseline at Day 112 (EOS): number analyzed (Participants) | 22 | 39 | 33
  Change from Baseline at Day 112 (EOS) | -1.26 (3.014) | -1.66 (3.543) | 0.35 (2.125)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 28; Test type: Other — Change from baseline was analyzed using a repeated measures model which included effects for treatment, visit, treatment by visit interaction, stratification factor (BMI group), baseline and baseline by visit interaction. BMI was separated into two groups, low BMI (Asian<30 and Non-Asian<35) and high BMI (Asian >=30 and Non-Asian>=35); p = 0.8402, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.079, 90% CI 2-sided [-0.724 to 0.567], Standard Error of Mean 0.389
Statistical Analysis 2: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 42; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.7607, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.144, 90% CI 2-sided [-0.927 to 0.639], Standard Error of Mean 0.472
Statistical Analysis 3: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 56; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.6406, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.228, 90% CI 2-sided [-1.037 to 0.581], Standard Error of Mean 0.487
Statistical Analysis 4: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 84; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.8185, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.158, 90% CI 2-sided [-1.294 to 0.979], Standard Error of Mean 0.685
Statistical Analysis 5: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 112 (EOS); Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.7804, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.214, 90% CI 2-sided [-1.485 to 1.057], Standard Error of Mean 0.766
Statistical Analysis 6: Comparison: LMB763 100 mg vs Pooled Placebo; Day 28; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.1403, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.598, 90% CI 2-sided [-1.265 to 0.070], Standard Error of Mean 0.402
Statistical Analysis 7: Comparison: LMB763 100 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0603, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.930, 90% CI 2-sided [-1.743 to -0.117], Standard Error of Mean 0.490
Statistical Analysis 8: Comparison: LMB763 100 mg vs Pooled Placebo; Day 56; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0090, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -1.344, 90% CI 2-sided [-2.182 to -0.506], Standard Error of Mean 0.505
Statistical Analysis 9: Comparison: LMB763 100 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0134, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -1.787, 90% CI 2-sided [-2.965 to -0.609], Standard Error of Mean 0.710
Statistical Analysis 10: Comparison: LMB763 100 mg vs Pooled Placebo; Day 112 (EOS); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0087, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -2.123, 90% CI 2-sided [-3.439 to -0.807], Standard Error of Mean 0.793
Statistical Analysis 11: Comparison: LMB763 50 mg vs Pooled Placebo; Day 28; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.1609, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.519, 90% CI 2-sided [-1.130 to 0.091], Standard Error of Mean 0.368
Statistical Analysis 12: Comparison: LMB763 50 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0797, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.786, 90% CI 2-sided [-1.524 to -0.049], Standard Error of Mean 0.444
Statistical Analysis 13: Comparison: LMB763 50 mg vs Pooled Placebo; Day 56; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0159, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -1.116, 90% CI 2-sided [-1.872 to -0.360], Standard Error of Mean 0.455
Statistical Analysis 14: Comparison: LMB763 50 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0118, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -1.630, 90% CI 2-sided [-2.684 to -0.575], Standard Error of Mean 0.635
Statistical Analysis 15: Comparison: LMB763 50 mg vs Pooled Placebo; Day 112 (EOS); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0076, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -1.909, 90% CI 2-sided [-3.072 to -0.746], Standard Error of Mean 0.700

9. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Baseline was defined as the last available measurement prior to the first dose at specified visit (day).
Time Frame: Baseline to Days 28, 42, 56, 84 and 112 (EOS)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)
Groups:
- Pooled Placebo: LMB763 100 mg or 50 mg matching placebo was self-administered orally once daily for 12 weeks (84 days) under fasted conditions (no food or drink for at least 6 hours).
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
kilograms per meter square (kg/m^2)
  Baseline for Day 28 Analysis: number analyzed (Participants) | 30 | 43 | 37
  Baseline for Day 28 Analysis | 34.81 (5.641) | 34.41 (5.270) | 34.93 (5.180)
  Change from Baseline at Day 28: number analyzed (Participants) | 30 | 43 | 37
  Change from Baseline at Day 28 | -0.29 (0.545) | -0.26 (0.638) | -0.05 (0.511)
  Baseline for Day 42 Analysis: number analyzed (Participants) | 27 | 43 | 34
  Baseline for Day 42 Analysis | 34.05 (5.162) | 34.41 (5.270) | 34.56 (5.233)
  Change from Baseline at Day 42: number analyzed (Participants) | 27 | 43 | 34
  Change from Baseline at Day 42 | -0.36 (0.591) | -0.40 (0.845) | -0.08 (0.572)
  Baseline for Day 56 Analysis: number analyzed (Participants) | 26 | 42 | 35
  Baseline for Day 56 Analysis | 34.12 (5.253) | 34.37 (5.327) | 34.75 (5.269)
  Change from Baseline at Day 56: number analyzed (Participants) | 26 | 42 | 35
  Change from Baseline at Day 56 | -0.50 (0.688) | -0.49 (0.799) | -0.10 (0.663)
  Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 40 | 34
  Baseline for Day 84 Analysis | 34.18 (5.467) | 34.04 (5.190) | 34.89 (5.275)
  Change from Baseline at Day 84: number analyzed (Participants) | 24 | 40 | 34
  Change from Baseline at Day 84 | -0.52 (0.764) | -0.72 (1.215) | -0.09 (0.718)
  Baseline for Day 112 (EOS) Analysis: number analyzed (Participants) | 22 | 39 | 33
  Baseline for Day 112 (EOS) Analysis | 34.60 (5.522) | 33.82 (4.980) | 34.96 (5.342)
  Change from Baseline at Day 112 (EOS): number analyzed (Participants) | 22 | 39 | 33
  Change from Baseline at Day 112 (EOS) | -0.45 (0.974) | -0.60 (1.276) | 0.12 (0.776)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 28; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.8127, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.033, 90% CI 2-sided [-0.260 to 0.195], Standard Error of Mean 0.137
Statistical Analysis 2: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 42; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.8901, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.023, 90% CI 2-sided [-0.298 to 0.252], Standard Error of Mean 0.166
Statistical Analysis 3: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 56; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.6209, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.088, 90% CI 2-sided [-0.381 to 0.205], Standard Error of Mean 0.177
Statistical Analysis 4: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 84; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.8398, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.048, 90% CI 2-sided [-0.444 to 0.347], Standard Error of Mean 0.238
Statistical Analysis 5: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 112 (EOS); Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.7839, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.073, 90% CI 2-sided [-0.515 to 0.369], Standard Error of Mean 0.266
Statistical Analysis 6: Comparison: LMB763 100 mg vs Pooled Placebo; Day 28; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0911, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.241, 90% CI 2-sided [-0.476 to -0.006], Standard Error of Mean 0.141
Statistical Analysis 7: Comparison: LMB763 100 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0520, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.338, 90% CI 2-sided [-0.623 to -0.053], Standard Error of Mean 0.172
Statistical Analysis 8: Comparison: LMB763 100 mg vs Pooled Placebo; Day 56; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0085, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.490, 90% CI 2-sided [-0.793 to -0.187], Standard Error of Mean 0.183
Statistical Analysis 9: Comparison: LMB763 100 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0091, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.657, 90% CI 2-sided [-1.067 to -0.247], Standard Error of Mean 0.247
Statistical Analysis 10: Comparison: LMB763 100 mg vs Pooled Placebo; Day 112 (EOS); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0070, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.759, 90% CI 2-sided [-1.216 to -0.302], Standard Error of Mean 0.275
Statistical Analysis 11: Comparison: LMB763 50 mg vs Pooled Placebo; Day 28; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.1092, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.208, 90% CI 2-sided [-0.423 to 0.006], Standard Error of Mean 0.129
Statistical Analysis 12: Comparison: LMB763 50 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0457, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.315, 90% CI 2-sided [-0.574 to -0.056], Standard Error of Mean 0.156
Statistical Analysis 13: Comparison: LMB763 50 mg vs Pooled Placebo; Day 56; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0162, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.402, 90% CI 2-sided [-0.676 to -0.129], Standard Error of Mean 0.165
Statistical Analysis 14: Comparison: LMB763 50 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0070, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.608, 90% CI 2-sided [-0.975 to -0.242], Standard Error of Mean 0.221
Statistical Analysis 15: Comparison: LMB763 50 mg vs Pooled Placebo; Day 112 (EOS); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0060, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.686, 90% CI 2-sided [-1.091 to -0.281], Standard Error of Mean 0.244

10. Secondary Outcome: Change From Baseline in Waist to Hip Ratio
Description: Baseline was defined as the last available measurement prior to the first dose.
Time Frame: Baseline to Days 28, 42, 56, 84 and 112 (EOS)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
ratio
  Baseline for Day 28 Analysis: number analyzed (Participants) | 30 | 43 | 36
  Baseline for Day 28 Analysis | 0.96 (0.065) | 0.96 (0.055) | 0.95 (0.089)
  Change from Baseline at Day 28: number analyzed (Participants) | 30 | 43 | 36
  Change from Baseline at Day 28 | 0.00 (0.039) | 0.00 (0.034) | -0.00 (0.039)
  Baseline for Day 42 Analysis: number analyzed (Participants) | 27 | 40 | 34
  Baseline for Day 42 Analysis | 0.96 (0.061) | 0.95 (0.056) | 0.96 (0.086)
  Change from Baseline at Day 42: number analyzed (Participants) | 27 | 40 | 34
  Change from Baseline at Day 42 | 0.01 (0.077) | -0.00 (0.039) | 0.00 (0.036)
  Baseline for Day 56 Analysis: number analyzed (Participants) | 25 | 42 | 34
  Baseline for Day 56 Analysis | 0.96 (0.061) | 0.96 (0.054) | 0.96 (0.087)
  Change from Baseline at Day 56: number analyzed (Participants) | 25 | 42 | 34
  Change from Baseline at Day 56 | -0.00 (0.029) | -0.00 (0.033) | -0.01 (0.029)
  Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 40 | 34
  Baseline for Day 84 Analysis | 0.95 (0.063) | 0.96 (0.055) | 0.96 (0.087)
  Change from Baseline at Day 84: number analyzed (Participants) | 24 | 40 | 34
  Change from Baseline at Day 84 | 0.00 (0.043) | -0.01 (0.044) | 0.01 (0.046)
  Baseline for Day 112 (EOS) Analysis: number analyzed (Participants) | 22 | 39 | 33
  Baseline for Day 112 (EOS) Analysis | 0.96 (0.059) | 0.96 (0.054) | 0.96 (0.087)
  Change from Baseline at Day 112 (EOS): number analyzed (Participants) | 22 | 39 | 33
  Change from Baseline at Day 112 (EOS) | -0.00 (0.030) | 0.00 (0.050) | -0.00 (0.037)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 28; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.9927, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.000, 90% CI 2-sided [-0.015 to 0.014], Standard Error of Mean 0.009
Statistical Analysis 2: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 42; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.2794, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.014, 90% CI 2-sided [-0.007 to 0.035], Standard Error of Mean 0.013
Statistical Analysis 3: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 56; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.9032, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.001, 90% CI 2-sided [-0.012 to 0.013], Standard Error of Mean 0.007
Statistical Analysis 4: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 84; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.4163, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.009, 90% CI 2-sided [-0.009 to 0.027], Standard Error of Mean 0.011
Statistical Analysis 5: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 112 (EOS); Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.7001, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.004, 90% CI 2-sided [-0.022 to 0.014], Standard Error of Mean 0.011
Statistical Analysis 6: Comparison: LMB763 100 mg vs Pooled Placebo; Day 28; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.5367, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.006, 90% CI 2-sided [-0.009 to 0.021], Standard Error of Mean 0.009
Statistical Analysis 7: Comparison: LMB763 100 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.5496, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.008, 90% CI 2-sided [-0.014 to 0.030], Standard Error of Mean 0.013
Statistical Analysis 8: Comparison: LMB763 100 mg vs Pooled Placebo; Day 56; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.6844, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.003, 90% CI 2-sided [-0.010 to 0.016], Standard Error of Mean 0.008
Statistical Analysis 9: Comparison: LMB763 100 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.5695, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.007, 90% CI 2-sided [-0.025 to 0.012], Standard Error of Mean 0.011
Statistical Analysis 10: Comparison: LMB763 100 mg vs Pooled Placebo; Day 112 (EOS); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.8015, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.003, 90% CI 2-sided [-0.021 to 0.016], Standard Error of Mean 0.011
Statistical Analysis 11: Comparison: LMB763 50 mg vs Pooled Placebo; Day 28; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.4923, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.006, 90% CI 2-sided [-0.008 to 0.020], Standard Error of Mean 0.008
Statistical Analysis 12: Comparison: LMB763 50 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.6200, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.006, 90% CI 2-sided [-0.025 to 0.014], Standard Error of Mean 0.012
Statistical Analysis 13: Comparison: LMB763 50 mg vs Pooled Placebo; Day 56; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.7423, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.002, 90% CI 2-sided [-0.009 to 0.014], Standard Error of Mean 0.007
Statistical Analysis 14: Comparison: LMB763 50 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.1272, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = -0.016, 90% CI 2-sided [-0.032 to 0.001], Standard Error of Mean 0.010
Statistical Analysis 15: Comparison: LMB763 50 mg vs Pooled Placebo; Day 112 (EOS); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.8883, ANCOVA; An unstructured variance-covariance structure was used; Mean Difference (Final Values) = 0.001, 90% CI 2-sided [-0.015 to 0.017], Standard Error of Mean 0.010

11. Secondary Outcome: Change From to Baseline in Liver Stiffness
Description: Fibroscan® was performed where available to assess liver stiffness. Baseline was defined as the last available measurement prior to the first dose. Geometric Mean and Geometric Coefficient of Variation for change are based on log-transformed ratio to baseline (i.e., change from baseline in the log domain).
Time Frame: Baseline to Day 84 (Week 12)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kilopascal (kPa)
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 10 | 17 | 18
kilopascal (kPa)
  Baseline for Day 84 Analysis: number analyzed (Participants) | 7 | 15 | 16
  Baseline for Day 84 Analysis | 7.689 (71.1) | 6.082 (29.5) | 7.108 (52.5)
  Change from Baseline at Day 84: number analyzed (Participants) | 7 | 15 | 16
  Change from Baseline at Day 84 | 0.955 (35.3) | 1.053 (26.9) | 1.041 (38.6)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.9514, ANCOVA; Geometric Mean Ratios = 1.01, 90% CI 2-sided [0.84 to 1.21]
Statistical Analysis 2: Comparison: LMB763 100 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.5168, ANCOVA; Geometric Mean Ratios = 0.93, 90% CI 2-sided [0.78 to 1.12]
Statistical Analysis 3: Comparison: LMB763 50 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.3740, ANCOVA; Geometric Mean Ratios = 0.93, 90% CI 2-sided [0.80 to 1.07]

12. Secondary Outcome: Change From Baseline in Enhanced Liver Fibrosis (ELF) Test Panel
Description: The ADVIA CentaurR systems' ELF™ test is an in vitro diagnostic multivariate index assay that provides a single score by combining quantitative measurements of hyaluronic acid (HA), amino-terminal propeptide of type III procollagen (PIIINP), and tissue inhibitor of metalloproteinase 1 (TIMP-1) in human serum using the ADVIA Centaur XP, ADVIA Centaur XPT, and ADVIA Centaur CP systems in an algorithm. ELF score for the ADVIA Centaur systems is calculated by, first obtaining results for the ADVIA Centaur HA, PIIINP, and TIMP-1 assays and then using the following equation/algorithm:
  ADVIA Centaur XP/XPT:
  ELF score = 2.278 + 0.851 ln(CHA) + 0.751 ln(CP3NP) + 0.394 ln(CTIMP1)
  ADVIA Centaur CP:
  ELF score = 2.494 + 0.846 ln(CHA) + 0.735 ln(CP3NP) + 0.391 ln(CTIMP1) Concentrations (C) of each assay are in ng/mL
  Interpretation of ELF score is as follows:
  < 7.7 None to mild
  * 7.7 to < 9.8 Moderate
  * 9.8 Severe
Time Frame: Baseline to Days 42 and 84
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ELF score
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
ELF score
  Baseline for Day 42 Analysis: number analyzed (Participants) | 26 | 42 | 33
  Baseline for Day 42 Analysis | 9.063 (7.3) | 8.731 (8.2) | 9.212 (8.0)
  Change from Baseline at Day 42: number analyzed (Participants) | 26 | 42 | 33
  Change from Baseline at Day 42 | 1.005 (5.5) | 1.016 (5.8) | 1.009 (7.5)
  Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 37 | 33
  Baseline for Day 84 Analysis | 9.051 (7.7) | 8.739 (8.4) | 9.220 (7.8)
  Change from Baseline at Day 84: number analyzed (Participants) | 24 | 37 | 33
  Change from Baseline at Day 84 | 1.005 (5.9) | 1.030 (6.2) | 1.007 (6.3)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 42; Test type: Other — Log transformed ratio to baseline was analyzed using a repeated measures model which included effects for treatment, visit, treatment by visit interaction, stratification factor (BMI group), log-transformed baseline and log-transformed baseline by visit interaction. BMI was separated into two groups, low BMI (Asian<30 and Non-Asian<35) and high BMI (Asian >=30 and Non-Asian>=35); p = 0.9453, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.00, 90% CI 2-sided [0.97 to 1.02]
Statistical Analysis 2: Comparison: LMB763 100 mg vs LMB763 50 mg; Day 84; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.4344, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.99, 90% CI 2-sided [0.96 to 1.01]
Statistical Analysis 3: Comparison: LMB763 100 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.6390, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.99, 90% CI 2-sided [0.97 to 1.02]
Statistical Analysis 4: Comparison: LMB763 100 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.6329, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.99, 90% CI 2-sided [0.97 to 1.02]
Statistical Analysis 5: Comparison: LMB763 50 mg vs Pooled Placebo; Day 42; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.6640, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.99, 90% CI 2-sided [0.97 to 1.02]
Statistical Analysis 6: Comparison: LMB763 50 mg vs Pooled Placebo; Day 84; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.7517, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.00, 90% CI 2-sided [0.98 to 1.03]

13. Secondary Outcome: Change From Baseline in Fibrosis Biomarker Test
Description: Fibrosis Biomarker test included hyaluronic acid (HA), amino-terminal pro-peptide of procollagen type III (PIIINP), and tissue inhibitor of metalloproteinases (TIMP-1) as markers of liver fibrosis. Baseline was defined as the last available measurement prior to the first dose. Geometric Mean and Geometric Coefficient of Variation for change are based on log-transformed ratio to baseline (i.e., change from baseline in the log domain).
Time Frame: Baseline to Days 42 and 84
Population: PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. Number analyzed in the number of participants with all observations non-missing, including censored data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per liter (ug/L)
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
micrograms per liter (ug/L)
  HA: Baseline for Day 42 Analysis: number analyzed (Participants) | 26 | 43 | 33
  HA: Baseline for Day 42 Analysis | 33.646 (72.2) | 26.869 (75.4) | 39.282 (74.9)
  HA: Change from Baseline at Day 42: number analyzed (Participants) | 26 | 43 | 33
  HA: Change from Baseline at Day 42 | 1.002 (49.5) | 1.133 (54.4) | 1.111 (77.0)
  HA: Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 38 | 33
  HA: Baseline for Day 84 Analysis | 32.246 (72.9) | 27.320 (78.2) | 40.865 (79.5)
  HA: Change from Baseline at Day 84: number analyzed (Participants) | 24 | 38 | 33
  HA: Change from Baseline at Day 84 | 1.023 (54.0) | 1.254 (51.4) | 1.071 (64.9)
  PIIINP: Baseline for Day 42 Analysis: number analyzed (Participants) | 26 | 43 | 33
  PIIINP: Baseline for Day 42 Analysis | 9.023 (31.3) | 7.850 (28.2) | 9.087 (35.5)
  PIIINP: Change from Baseline at Day 42: number analyzed (Participants) | 26 | 43 | 33
  PIIINP: Change from Baseline at Day 42 | 1.016 (22.8) | 1.071 (24.3) | 1.010 (26.4)
  PIIINP: Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 38 | 33
  PIIINP: Baseline for Day 84 Analysis | 9.263 (34.6) | 7.859 (27.4) | 8.934 (32.3)
  PIIINP: Change from Baseline at Day 84: number analyzed (Participants) | 24 | 38 | 33
  PIIINP: Change from Baseline at Day 84 | 1.003 (21.2) | 1.048 (26.9) | 1.004 (20.1)
  TIMP-1: Baseline for Day 42 Analysis: number analyzed (Participants) | 26 | 43 | 33
  TIMP-1: Baseline for Day 42 Analysis | 242.99 (17.5) | 199.21 (78.4) | 254.37 (23.1)
  TIMP-1: Change from Baseline at Day 42: number analyzed (Participants) | 26 | 43 | 33
  TIMP-1: Change from Baseline at Day 42 | 1.060 (14.6) | 1.017 (11.9) | 0.995 (13.3)
  TIMP-1: Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 38 | 33
  TIMP-1: Baseline for Day 84 Analysis | 247.42 (18.8) | 193.32 (83.6) | 245.09 (20.5)
  TIMP-1: Change from Baseline at Day 84: number analyzed (Participants) | 24 | 38 | 33
  TIMP-1: Change from Baseline at Day 84 | 1.073 (17.0) | 1.036 (10.4) | 1.000 (19.2)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; HA: Day 42; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.7390, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.77 to 1.19]
Statistical Analysis 2: Comparison: LMB763 100 mg vs LMB763 50 mg; HA: Day 84; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.3086, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.88, 90% CI 2-sided [0.72 to 1.08]
Statistical Analysis 3: Comparison: LMB763 100 mg vs Pooled Placebo; HA: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.2880, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.86, 90% CI 2-sided [0.69 to 1.08]
Statistical Analysis 4: Comparison: LMB763 100 mg vs Pooled Placebo; HA: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.4446, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.91, 90% CI 2-sided [0.73 to 1.12]
Statistical Analysis 5: Comparison: LMB763 50 mg vs Pooled Placebo; HA: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.4127, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.90, 90% CI 2-sided [0.73 to 1.11]
Statistical Analysis 6: Comparison: LMB763 50 mg vs Pooled Placebo; HA: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.8074, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.03, 90% CI 2-sided [0.85 to 1.25]
Statistical Analysis 7: Comparison: LMB763 100 mg vs LMB763 50 mg; PIIINP: Day 42; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.6935, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.98, 90% CI 2-sided [0.88 to 1.08]
Statistical Analysis 8: Comparison: LMB763 100 mg vs LMB763 50 mg; PIIINP: Day 84; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.9145, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.99, 90% CI 2-sided [0.90 to 1.09]
Statistical Analysis 9: Comparison: LMB763 100 mg vs Pooled Placebo; PIIINP: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.9131, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.01, 90% CI 2-sided [0.91 to 1.12]
Statistical Analysis 10: Comparison: LMB763 100 mg vs Pooled Placebo; PIIINP: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.9988, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.00, 90% CI 2-sided [0.91 to 1.10]
Statistical Analysis 11: Comparison: LMB763 50 mg vs Pooled Placebo; PIIINP: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.5873, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.03, 90% CI 2-sided [0.94 to 1.13]
Statistical Analysis 12: Comparison: LMB763 50 mg vs Pooled Placebo; PIIINP: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.9050, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.01, 90% CI 2-sided [0.92 to 1.10]
Statistical Analysis 13: Comparison: LMB763 100 mg vs LMB763 50 mg; TIMP-1: Day 42; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.1458, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.05, 90% CI 2-sided [0.99 to 1.11]
Statistical Analysis 14: Comparison: LMB763 100 mg vs LMB763 50 mg; TIMP-1: Day 84; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.2048, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.05, 90% CI 2-sided [0.98 to 1.12]
Statistical Analysis 15: Comparison: LMB763 100 mg vs Pooled Placebo; TIMP-1: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1051, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.06, 90% CI 2-sided [1.00 to 1.12]
Statistical Analysis 16: Comparison: LMB763 100 mg vs Pooled Placebo; TIMP-1: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0717, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.08, 90% CI 2-sided [1.01 to 1.15]
Statistical Analysis 17: Comparison: LMB763 50 mg vs Pooled Placebo; TIMP-1: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.8083, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.01, 90% CI 2-sided [0.96 to 1.06]
Statistical Analysis 18: Comparison: LMB763 50 mg vs Pooled Placebo; TIMP-1: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.5361, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.02, 90% CI 2-sided [0.96 to 1.09]

14. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Cholesterol (Chol) and Triglycerides (TG)
Description: Lipid measurements were collected under fasted conditions. Baseline was defined as the last available measurement prior to the first dose. Geometric Mean and Geometric Coefficient of Variation for change are based on log-transformed ratio to baseline (i.e., change from baseline in the log domain).
Time Frame: Baseline to Days 7, 14, 28, 42, 56, 84 and 112 (EOS)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per deciliter (mg/dL)
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
milligrams per deciliter (mg/dL)
  Chol: Baseline for Day 7 Analysis: number analyzed (Participants) | 36 | 44 | 40
  Chol: Baseline for Day 7 Analysis | 184.85 (23.0) | 183.30 (22.1) | 188.97 (22.0)
  Chol: Change from Baseline at Day 7: number analyzed (Participants) | 36 | 44 | 40
  Chol: Change from Baseline at Day 7 | 0.957 (14.5) | 1.001 (9.0) | 1.002 (10.2)
  Chol: Baseline for Day 14 Analysis: number analyzed (Participants) | 34 | 44 | 40
  Chol: Baseline for Day 14 Analysis | 186.57 (23.1) | 183.30 (22.1) | 188.97 (22.0)
  Chol: Change from Baseline at Day 14: number analyzed (Participants) | 34 | 44 | 40
  Chol: Change from Baseline at Day 14 | 0.963 (17.0) | 1.037 (11.8) | 1.000 (10.4)
  Chol: Baseline for Day 28 Analysis: number analyzed (Participants) | 29 | 43 | 37
  Chol: Baseline for Day 28 Analysis | 188.09 (23.2) | 183.50 (22.3) | 190.44 (22.4)
  Chol: Change from Baseline at Day 28: number analyzed (Participants) | 29 | 43 | 37
  Chol: Change from Baseline at Day 28 | 0.952 (15.2) | 1.025 (14.6) | 1.007 (12.2)
  Chol: Baseline for Day 42 Analysis: number analyzed (Participants) | 19 | 42 | 30
  Chol: Baseline for Day 42 Analysis | 206.50 (18.3) | 182.59 (22.3) | 191.65 (21.1)
  Chol: Change from Baseline at Day 42: number analyzed (Participants) | 19 | 42 | 30
  Chol: Change from Baseline at Day 42 | 0.943 (17.2) | 1.001 (15.1) | 0.940 (14.2)
  Chol: Baseline for Day 56 Analysis: number analyzed (Participants) | 25 | 41 | 33
  Chol: Baseline for Day 56 Analysis | 192.25 (22.5) | 182.39 (22.5) | 190.33 (21.0)
  Chol: Change from Baseline at Day 56: number analyzed (Participants) | 25 | 41 | 33
  Chol: Change from Baseline at Day 56 | 0.963 (17.2) | 1.033 (16.1) | 1.002 (15.2)
  Chol: Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 40 | 32
  Chol: Baseline for Day 84 Analysis | 188.88 (22.0) | 181.63 (22.4) | 187.20 (23.6)
  Chol: Change from Baseline at Day 84: number analyzed (Participants) | 24 | 40 | 32
  Chol: Change from Baseline at Day 84 | 0.958 (17.9) | 1.037 (18.9) | 1.006 (13.5)
  Chol: Baseline for Day 112 (EOS) Analysis: number analyzed (Participants) | 22 | 39 | 33
  Chol: Baseline for Day 112 (EOS) Analysis | 187.34 (22.8) | 181.47 (22.0) | 187.13 (23.1)
  Chol: Change from Baseline at Day 112 (EOS): number analyzed (Participants) | 22 | 39 | 33
  Chol: Change from Baseline at Day 112 (EOS) | 0.989 (13.6) | 1.039 (16.8) | 1.009 (13.2)
  TG: Baseline for Day 7 Analysis: number analyzed (Participants) | 36 | 44 | 40
  TG: Baseline for Day 7 Analysis | 185.66 (55.0) | 198.88 (47.8) | 175.18 (58.7)
  TG: Change from Baseline at Day 7: number analyzed (Participants) | 36 | 44 | 40
  TG: Change from Baseline at Day 7 | 0.876 (38.8) | 0.854 (25.8) | 1.020 (28.6)
  TG: Baseline for Day 14 Analysis: number analyzed (Participants) | 34 | 44 | 40
  TG: Baseline for Day 14 Analysis | 178.22 (50.5) | 198.88 (47.8) | 175.18 (58.7)
  TG: Change from Baseline at Day 14: number analyzed (Participants) | 34 | 44 | 40
  TG: Change from Baseline at Day 14 | 0.864 (36.2) | 0.881 (28.1) | 1.013 (35.9)
  TG: Baseline for Day 28 Analysis: number analyzed (Participants) | 29 | 43 | 37
  TG: Baseline for Day 28 Analysis | 166.54 (45.0) | 201.00 (47.7) | 177.66 (60.6)
  TG: Change from Baseline at Day 28: number analyzed (Participants) | 29 | 43 | 37
  TG: Change from Baseline at Day 28 | 0.968 (36.4) | 0.937 (37.0) | 0.971 (33.7)
  TG: Baseline for Day 42 Analysis: number analyzed (Participants) | 19 | 42 | 30
  TG: Baseline for Day 42 Analysis | 181.97 (44.6) | 203.65 (47.4) | 174.48 (64.4)
  TG: Change from Baseline at Day 42: number analyzed (Participants) | 19 | 42 | 30
  TG: Change from Baseline at Day 42 | 0.868 (34.5) | 0.872 (36.1) | 0.920 (35.2)
  TG: Baseline for Day 56 Analysis: number analyzed (Participants) | 25 | 41 | 33
  TG: Baseline for Day 56 Analysis | 167.66 (47.5) | 202.64 (48.8) | 174.78 (60.6)
  TG: Change from Baseline at Day 56: number analyzed (Participants) | 25 | 41 | 33
  TG: Change from Baseline at Day 56 | 0.932 (34.2) | 0.948 (38.9) | 0.965 (28.1)
  TG: Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 40 | 32
  TG: Baseline for Day 84 Analysis | 163.71 (48.6) | 201.96 (49.5) | 184.99 (59.7)
  TG: Change from Baseline at Day 84: number analyzed (Participants) | 24 | 40 | 32
  TG: Change from Baseline at Day 84 | 0.863 (43.8) | 0.956 (45.8) | 0.947 (33.3)
  TG: Baseline for Day 112 (EOS) Analysis: number analyzed (Participants) | 22 | 39 | 33
  TG: Baseline for Day 112 (EOS) Analysis | 172.80 (46.1) | 203.55 (49.2) | 179.36 (62.5)
  TG: Change from Baseline at Day 112 (EOS): number analyzed (Participants) | 22 | 39 | 33
  TG: Change from Baseline at Day 112 (EOS) | 0.931 (38.5) | 1.003 (39.9) | 1.039 (39.0)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Cholesterol: Day 7; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0858, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.92 to 1.00]
Statistical Analysis 2: Comparison: LMB763 100 mg vs LMB763 50 mg; Cholesterol: Day 14; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0096, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.93, 90% CI 2-sided [0.88 to 0.97]
Statistical Analysis 3: Comparison: LMB763 100 mg vs LMB763 50 mg; Cholesterol: Day 28; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0284, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.93, 90% CI 2-sided [0.88 to 0.98]
Statistical Analysis 4: Comparison: LMB763 100 mg vs LMB763 50 mg; Cholesterol: Day 42; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.1330, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.95, 90% CI 2-sided [0.89 to 1.01]
Statistical Analysis 5: Comparison: LMB763 100 mg vs LMB763 50 mg; Cholesterol: Day 56; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.2032, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.95, 90% CI 2-sided [0.89 to 1.01]
Statistical Analysis 6: Comparison: LMB763 100 mg vs LMB763 50 mg; Cholesterol: Day 84; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.1141, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.87 to 1.00]
Statistical Analysis 7: Comparison: LMB763 100 mg vs LMB763 50 mg; Cholesterol: Day 112 (EOS); Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.1342, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.88 to 1.01]
Statistical Analysis 8: Comparison: LMB763 100 mg vs Pooled Placebo; Cholesterol: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0771, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.92 to 1.00]
Statistical Analysis 9: Comparison: LMB763 100 mg vs Pooled Placebo; Cholesterol: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1510, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.91 to 1.01]
Statistical Analysis 10: Comparison: LMB763 100 mg vs Pooled Placebo; Cholesterol: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0744, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.89 to 1.00]
Statistical Analysis 11: Comparison: LMB763 100 mg vs Pooled Placebo; Cholesterol: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.8365, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.99, 90% CI 2-sided [0.93 to 1.06]
Statistical Analysis 12: Comparison: LMB763 100 mg vs Pooled Placebo; Cholesterol: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.6091, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.98, 90% CI 2-sided [0.92 to 1.05]
Statistical Analysis 13: Comparison: LMB763 100 mg vs Pooled Placebo; Cholesterol: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.3621, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.90 to 1.03]
Statistical Analysis 14: Comparison: LMB763 100 mg vs Pooled Placebo; Cholesterol: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.5031, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.97, 90% CI 2-sided [0.91 to 1.04]
Statistical Analysis 15: Comparison: LMB763 50 mg vs Pooled Placebo; Cholesterol: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.9244, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.00, 90% CI 2-sided [0.96 to 1.04]
Statistical Analysis 16: Comparison: LMB763 50 mg vs Pooled Placebo; Cholesterol: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.2360, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.03, 90% CI 2-sided [0.99 to 1.08]
Statistical Analysis 17: Comparison: LMB763 50 mg vs Pooled Placebo; Cholesterol: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.6990, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.01, 90% CI 2-sided [0.96 to 1.07]
Statistical Analysis 18: Comparison: LMB763 50 mg vs Pooled Placebo; Cholesterol: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1590, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.05, 90% CI 2-sided [0.99 to 1.11]
Statistical Analysis 19: Comparison: LMB763 50 mg vs Pooled Placebo; Cholesterol: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.4256, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.03, 90% CI 2-sided [0.97 to 1.09]
Statistical Analysis 20: Comparison: LMB763 50 mg vs Pooled Placebo; Cholesterol: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.4901, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.03, 90% CI 2-sided [0.96 to 1.09]
Statistical Analysis 21: Comparison: LMB763 50 mg vs Pooled Placebo; Cholesterol: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.3648, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.03, 90% CI 2-sided [0.97 to 1.09]
Statistical Analysis 22: Comparison: LMB763 100 mg vs LMB763 50 mg; Triglycerides: Day 7; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.8891, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.01, 90% CI 2-sided [0.91 to 1.12]
Statistical Analysis 23: Comparison: LMB763 100 mg vs LMB763 50 mg; Triglycerides: Day 14; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.4817, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.95, 90% CI 2-sided [0.85 to 1.07]
Statistical Analysis 24: Comparison: LMB763 100 mg vs LMB763 50 mg; Triglycerides: Day 28; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.6022, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.84 to 1.09]
Statistical Analysis 25: Comparison: LMB763 100 mg vs LMB763 50 mg; Triglycerides: Day 42; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.4470, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.83 to 1.07]
Statistical Analysis 26: Comparison: LMB763 100 mg vs LMB763 50 mg; Triglycerides: Day 56; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.4342, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.83 to 1.07]
Statistical Analysis 27: Comparison: LMB763 100 mg vs LMB763 50 mg; Triglycerides: Day 84; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0891, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.85, 90% CI 2-sided [0.73 to 0.99]
Statistical Analysis 28: Comparison: LMB763 100 mg vs LMB763 50 mg; Triglycerides: Day 112 (EOS); Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.2260, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.89, 90% CI 2-sided [0.77 to 1.04]
Statistical Analysis 29: Comparison: LMB763 100 mg vs Pooled Placebo; Triglycerides: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0324, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.87, 90% CI 2-sided [0.78 to 0.97]
Statistical Analysis 30: Comparison: LMB763 100 mg vs Pooled Placebo; Triglycerides: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0291, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.85, 90% CI 2-sided [0.76 to 0.96]
Statistical Analysis 31: Comparison: LMB763 100 mg vs Pooled Placebo; Triglycerides: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.5755, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.84 to 1.09]
Statistical Analysis 32: Comparison: LMB763 100 mg vs Pooled Placebo; Triglycerides: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.3070, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.92, 90% CI 2-sided [0.80 to 1.05]
Statistical Analysis 33: Comparison: LMB763 100 mg vs Pooled Placebo; Triglycerides: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.7752, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.98, 90% CI 2-sided [0.86 to 1.12]
Statistical Analysis 34: Comparison: LMB763 100 mg vs Pooled Placebo; Triglycerides: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1803, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.88, 90% CI 2-sided [0.75 to 1.03]
Statistical Analysis 35: Comparison: LMB763 100 mg vs Pooled Placebo; Triglycerides: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.2414, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.89, 90% CI 2-sided [0.76 to 1.05]
Statistical Analysis 36: Comparison: LMB763 50 mg vs Pooled Placebo; Triglycerides: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0179, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.86, 90% CI 2-sided [0.77 to 0.95]
Statistical Analysis 37: Comparison: LMB763 50 mg vs Pooled Placebo; Triglycerides: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1125, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.90, 90% CI 2-sided [0.80 to 1.00]
Statistical Analysis 38: Comparison: LMB763 50 mg vs Pooled Placebo; Triglycerides: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.9572, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.00, 90% CI 2-sided [0.88 to 1.12]
Statistical Analysis 39: Comparison: LMB763 50 mg vs Pooled Placebo; Triglycerides: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.7372, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.98, 90% CI 2-sided [0.87 to 1.10]
Statistical Analysis 40: Comparison: LMB763 50 mg vs Pooled Placebo; Triglycerides: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.6015, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.04, 90% CI 2-sided [0.92 to 1.17]
Statistical Analysis 41: Comparison: LMB763 50 mg vs Pooled Placebo; Triglycerides: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.7261, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.03, 90% CI 2-sided [0.89 to 1.19]
Statistical Analysis 42: Comparison: LMB763 50 mg vs Pooled Placebo; Triglycerides: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.9892, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.00, 90% CI 2-sided [0.87 to 1.15]

15. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: High-density Lipoprotein (HDL) and Low-density Lipoprotein (LDL) Cholesterol
Description: Baseline was defined as the last available measurement prior to the first dose. Geometric Mean and Geometric Coefficient of Variation for change are based on log-transformed ratio to baseline (i.e., change from baseline in the log domain).
Time Frame: Baseline to Days 7, 14, 28, 42, 56, 84 and 112 (EOS)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimole per liter (mmol/L)
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
millimole per liter (mmol/L)
  HDL: Baseline for Day 7 Analysis: number analyzed (Participants) | 36 | 44 | 40
  HDL: Baseline for Day 7 Analysis | 1.059 (30.0) | 1.014 (25.4) | 1.206 (28.2)
  HDL: Change from Baseline at Day 7: number analyzed (Participants) | 36 | 44 | 40
  HDL: Change from Baseline at Day 7 | 0.874 (15.0) | 0.969 (10.0) | 1.017 (12.7)
  HDL: Baseline for Day 14 Analysis: number analyzed (Participants) | 34 | 44 | 40
  HDL: Baseline for Day 14 Analysis | 1.093 (24.8) | 1.014 (25.4) | 1.206 (28.2)
  HDL: Change from Baseline at Day 14: number analyzed (Participants) | 34 | 44 | 40
  HDL: Change from Baseline at Day 14 | 0.876 (19.1) | 0.982 (13.4) | 0.979 (10.0)
  HDL: Baseline for Day 28 Analysis: number analyzed (Participants) | 29 | 43 | 37
  HDL: Baseline for Day 28 Analysis | 1.143 (23.8) | 1.014 (25.7) | 1.221 (28.9)
  HDL: Change from Baseline at Day 28: number analyzed (Participants) | 29 | 43 | 37
  HDL: Change from Baseline at Day 28 | 0.862 (14.1) | 0.952 (15.1) | 1.009 (14.7)
  HDL: Baseline for Day 42 Analysis: number analyzed (Participants) | 19 | 42 | 30
  HDL: Baseline for Day 42 Analysis | 1.172 (26.9) | 1.007 (25.7) | 1.212 (30.6)
  HDL: Change from Baseline at Day 42: number analyzed (Participants) | 19 | 42 | 30
  HDL: Change from Baseline at Day 42 | 0.888 (19.4) | 0.941 (15.5) | 1.005 (12.2)
  HDL: Baseline for Day 56 Analysis: number analyzed (Participants) | 24 | 41 | 33
  HDL: Baseline for Day 56 Analysis | 1.148 (25.5) | 1.008 (25.9) | 1.226 (29.1)
  HDL: Change from Baseline at Day 56: number analyzed (Participants) | 24 | 41 | 33
  HDL: Change from Baseline at Day 56 | 0.875 (17.0) | 0.956 (15.1) | 1.022 (13.9)
  HDL: Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 40 | 32
  HDL: Baseline for Day 84 Analysis | 1.158 (24.9) | 1.016 (26.6) | 1.219 (29.7)
  HDL: Change from Baseline at Day 84: number analyzed (Participants) | 24 | 40 | 32
  HDL: Change from Baseline at Day 84 | 0.891 (16.1) | 0.920 (19.9) | 1.031 (12.5)
  HDL: Baseline for Day 112 (EOS) Analysis: number analyzed (Participants) | 22 | 39 | 33
  HDL: Baseline for Day 112 (EOS) Analysis | 1.115 (22.1) | 1.013 (26.1) | 1.218 (29.6)
  HDL: Change from Baseline at Day 112 (EOS): number analyzed (Participants) | 22 | 39 | 33
  HDL: Change from Baseline at Day 112 (EOS) | 1.004 (14.5) | 1.037 (17.2) | 1.007 (11.5)
  LDL: Baseline for Day 7 Analysis: number analyzed (Participants) | 34 | 43 | 37
  LDL: Baseline for Day 7 Analysis | 2.647 (39.0) | 2.591 (40.6) | 2.628 (34.2)
  LDL: Change from Baseline at Day 7: number analyzed (Participants) | 34 | 43 | 37
  LDL: Change from Baseline at Day 7 | 1.009 (18.7) | 1.076 (20.2) | 0.977 (17.1)
  LDL: Baseline for Day 14 Analysis: number analyzed (Participants) | 33 | 43 | 35
  LDL: Baseline for Day 14 Analysis | 2.664 (39.8) | 2.591 (40.6) | 2.666 (34.3)
  LDL: Change from Baseline at Day 14: number analyzed (Participants) | 33 | 43 | 35
  LDL: Change from Baseline at Day 14 | 1.021 (23.6) | 1.125 (19.7) | 0.998 (14.3)
  LDL: Baseline for Day 28 Analysis: number analyzed (Participants) | 29 | 41 | 36
  LDL: Baseline for Day 28 Analysis | 2.612 (39.4) | 2.553 (40.7) | 2.614 (36.3)
  LDL: Change from Baseline at Day 28: number analyzed (Participants) | 29 | 41 | 36
  LDL: Change from Baseline at Day 28 | 0.996 (27.5) | 1.092 (23.0) | 1.017 (15.7)
  LDL: Baseline for Day 42 Analysis: number analyzed (Participants) | 19 | 41 | 28
  LDL: Baseline for Day 42 Analysis | 3.070 (28.7) | 2.559 (41.0) | 2.679 (35.1)
  LDL: Change from Baseline at Day 42: number analyzed (Participants) | 19 | 41 | 28
  LDL: Change from Baseline at Day 42 | 0.989 (29.9) | 1.079 (24.5) | 0.914 (21.1)
  LDL: Baseline for Day 56 Analysis: number analyzed (Participants) | 24 | 38 | 32
  LDL: Baseline for Day 56 Analysis | 2.841 (32.0) | 2.527 (42.0) | 2.621 (36.0)
  LDL: Change from Baseline at Day 56: number analyzed (Participants) | 24 | 38 | 32
  LDL: Change from Baseline at Day 56 | 1.011 (27.9) | 1.091 (24.8) | 0.991 (24.7)
  LDL: Baseline for Day 84 Analysis: number analyzed (Participants) | 24 | 38 | 29
  LDL: Baseline for Day 84 Analysis | 2.725 (30.8) | 2.528 (41.8) | 2.498 (36.8)
  LDL: Change from Baseline at Day 84: number analyzed (Participants) | 24 | 38 | 29
  LDL: Change from Baseline at Day 84 | 1.029 (22.5) | 1.107 (31.7) | 1.025 (22.2)
  LDL: Baseline for Day 112 (EOS) Analysis: number analyzed (Participants) | 22 | 35 | 29
  LDL: Baseline for Day 112 (EOS) Analysis | 2.695 (31.6) | 2.418 (40.0) | 2.482 (36.2)
  LDL: Change from Baseline at Day 112 (EOS): number analyzed (Participants) | 22 | 35 | 29
  LDL: Change from Baseline at Day 112 (EOS) | 1.010 (18.7) | 1.035 (34.1) | 1.026 (19.9)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; HDL Cholesterol: Day 7; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0005, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.91, 90% CI 2-sided [0.87 to 0.95]
Statistical Analysis 2: Comparison: LMB763 100 mg vs LMB763 50 mg; HDL Cholesterol: Day 14; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0005, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.89, 90% CI 2-sided [0.84 to 0.94]
Statistical Analysis 3: Comparison: LMB763 100 mg vs LMB763 50 mg; HDL Cholesterol: Day 28; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0062, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.91, 90% CI 2-sided [0.86 to 0.96]
Statistical Analysis 4: Comparison: LMB763 100 mg vs LMB763 50 mg; HDL Cholesterol: Day 42; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.1214, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.89 to 1.00]
Statistical Analysis 5: Comparison: LMB763 100 mg vs LMB763 50 mg; HDL Cholesterol: Day 56; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0043, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.90, 90% CI 2-sided [0.84 to 0.95]
Statistical Analysis 6: Comparison: LMB763 100 mg vs LMB763 50 mg; HDL Cholesterol: Day 84; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.2615, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.95, 90% CI 2-sided [0.89 to 1.02]
Statistical Analysis 7: Comparison: LMB763 100 mg vs LMB763 50 mg; HDL Cholesterol: Day 112 (EOS); Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.1331, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.88 to 1.01]
Statistical Analysis 8: Comparison: LMB763 100 mg vs Pooled Placebo; HDL Cholesterol: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p < .0001, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.85, 90% CI 2-sided [0.81 to 0.89]
Statistical Analysis 9: Comparison: LMB763 100 mg vs Pooled Placebo; HDL Cholesterol: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0001, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.88, 90% CI 2-sided [0.83 to 0.93]
Statistical Analysis 10: Comparison: LMB763 100 mg vs Pooled Placebo; HDL Cholesterol: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p < .0001, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.83, 90% CI 2-sided [0.79 to 0.88]
Statistical Analysis 11: Comparison: LMB763 100 mg vs Pooled Placebo; HDL Cholesterol: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0002, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.86, 90% CI 2-sided [0.81 to 0.92]
Statistical Analysis 12: Comparison: LMB763 100 mg vs Pooled Placebo; HDL Cholesterol: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p < .0001, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.82, 90% CI 2-sided [0.77 to 0.88]
Statistical Analysis 13: Comparison: LMB763 100 mg vs Pooled Placebo; HDL Cholesterol: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0002, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.84, 90% CI 2-sided [0.78 to 0.90]
Statistical Analysis 14: Comparison: LMB763 100 mg vs Pooled Placebo; HDL Cholesterol: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.2280, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.95, 90% CI 2-sided [0.89 to 1.02]
Statistical Analysis 15: Comparison: LMB763 50 mg vs Pooled Placebo; HDL Cholesterol: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0090, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.93, 90% CI 2-sided [0.89 to 0.97]
Statistical Analysis 16: Comparison: LMB763 50 mg vs Pooled Placebo; HDL Cholesterol: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.6237, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.98, 90% CI 2-sided [0.93 to 1.04]
Statistical Analysis 17: Comparison: LMB763 50 mg vs Pooled Placebo; HDL Cholesterol: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0080, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.91, 90% CI 2-sided [0.87 to 0.97]
Statistical Analysis 18: Comparison: LMB763 50 mg vs Pooled Placebo; HDL Cholesterol: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0105, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.91, 90% CI 2-sided [0.86 to 0.97]
Statistical Analysis 19: Comparison: LMB763 50 mg vs Pooled Placebo; HDL Cholesterol: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0217, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.92, 90% CI 2-sided [0.86 to 0.98]
Statistical Analysis 20: Comparison: LMB763 50 mg vs Pooled Placebo; HDL Cholesterol: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0031, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.88, 90% CI 2-sided [0.82 to 0.94]
Statistical Analysis 21: Comparison: LMB763 50 mg vs Pooled Placebo; HDL Cholesterol: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.7740, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.01, 90% CI 2-sided [0.95 to 1.07]
Statistical Analysis 22: Comparison: LMB763 100 mg vs LMB763 50 mg; LDL Cholesterol Friedwald: Day 7; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.1783, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.95, 90% CI 2-sided [0.89 to 1.01]
Statistical Analysis 23: Comparison: LMB763 100 mg vs LMB763 50 mg; LDL Cholesterol Friedwald: Day 14; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0219, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.91, 90% CI 2-sided [0.84 to 0.97]
Statistical Analysis 24: Comparison: LMB763 100 mg vs LMB763 50 mg; LDL Cholesterol Friedwald: Day 28; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.0719, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.92, 90% CI 2-sided [0.85 to 0.99]
Statistical Analysis 25: Comparison: LMB763 100 mg vs LMB763 50 mg; LDL Cholesterol Friedwald: Day 42; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.2199, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.93, 90% CI 2-sided [0.85 to 1.02]
Statistical Analysis 26: Comparison: LMB763 100 mg vs LMB763 50 mg; LDL Cholesterol Friedwald: Day 56; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.4928, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.96, 90% CI 2-sided [0.87 to 1.06]
Statistical Analysis 27: Comparison: LMB763 100 mg vs LMB763 50 mg; LDL Cholesterol Friedwald: Day 84; Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.3419, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.94, 90% CI 2-sided [0.85 to 1.05]
Statistical Analysis 28: Comparison: LMB763 100 mg vs LMB763 50 mg; LDL Cholesterol Friedwald: Day 112 (EOS); Test type: Other — [test comment as in outcome 2, analysis 2]; p = 0.7281, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.98, 90% CI 2-sided [0.88 to 1.09]
Statistical Analysis 29: Comparison: LMB763 100 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.3180, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.04, 90% CI 2-sided [0.97 to 1.12]
Statistical Analysis 30: Comparison: LMB763 100 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.6576, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.02, 90% CI 2-sided [0.95 to 1.10]
Statistical Analysis 31: Comparison: LMB763 100 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.6035, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 0.97, 90% CI 2-sided [0.90 to 1.06]
Statistical Analysis 32: Comparison: LMB763 100 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.3261, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.06, 90% CI 2-sided [0.96 to 1.17]
Statistical Analysis 33: Comparison: LMB763 100 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.5246, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.04, 90% CI 2-sided [0.94 to 1.15]
Statistical Analysis 34: Comparison: LMB763 100 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.7519, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.02, 90% CI 2-sided [0.92 to 1.14]
Statistical Analysis 35: Comparison: LMB763 100 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.9577, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.00, 90% CI 2-sided [0.89 to 1.12]
Statistical Analysis 36: Comparison: LMB763 50 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 7; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0160, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.10, 90% CI 2-sided [1.03 to 1.18]
Statistical Analysis 37: Comparison: LMB763 50 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0052, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.13, 90% CI 2-sided [1.05 to 1.21]
Statistical Analysis 38: Comparison: LMB763 50 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 28; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1822, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.06, 90% CI 2-sided [0.99 to 1.15]
Statistical Analysis 39: Comparison: LMB763 50 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 42; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.0159, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.14, 90% CI 2-sided [1.04 to 1.24]
Statistical Analysis 40: Comparison: LMB763 50 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 56; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1524, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.08, 90% CI 2-sided [0.99 to 1.19]
Statistical Analysis 41: Comparison: LMB763 50 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 84; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.1749, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.08, 90% CI 2-sided [0.98 to 1.20]
Statistical Analysis 42: Comparison: LMB763 50 mg vs Pooled Placebo; LDL Cholesterol Friedwald: Day 112 (EOS); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.7503, ANCOVA; An unstructured variance-covariance structure was used; Geometric Mean Ratios = 1.02, 90% CI 2-sided [0.92 to 1.13]

16. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) for Itching of Skin
Description: A 10 cm VAS was used to assess the severity of participants itch (ranging from 0 = no itch at all to 10 = the worst imaginable itch). The score (distance from left) on the VAS was recorded by the participant marking with a line and used to test for an effect of LMB763 over placebo. Baseline was defined as the last available measurement prior to the first dose. A positive change from Baseline indicates improvement.
Time Frame: Baseline to Day 84 (Week 12)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
Number analyzed (Participants) | 37 | 44 | 40
score on a scale
  Baseline for Day 84 Analysis: number analyzed (Participants) | 23 | 39 | 34
  Baseline for Day 84 Analysis | 8.87 (19.108) | 4.62 (10.356) | 9.68 (19.552)
  Change from Baseline at Day 84: number analyzed (Participants) | 23 | 39 | 34
  Change from Baseline at Day 84 | 9.35 (18.746) | 4.85 (21.798) | 2.03 (24.037)
Statistical Analysis 1: Comparison: LMB763 100 mg vs LMB763 50 mg; Test type: Other — Change from baseline was analyzed using an ANCOVA model which included effects for treatment, baseline and stratification factor (BMI group). BMI was separated into two groups, low BMI (Asian<30 and Non-Asian<35) and high BMI (Asian >=30 and Non-Asian>=35); p = 0.2073, ANCOVA; Mean Difference (Final Values) = 7.01, 90% CI 2-sided [-2.161 to 16.178], Standard Error of Mean 5.52
Statistical Analysis 2: Comparison: LMB763 100 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.2014, ANCOVA; Mean Difference (Final Values) = 7.23, 90% CI 2-sided [-2.106 to 16.563], Standard Error of Mean 5.62
Statistical Analysis 3: Comparison: LMB763 50 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.9645, ANCOVA; Mean Difference (Final Values) = 0.22, 90% CI 2-sided [-7.974 to 8.414], Standard Error of Mean 4.93

ADVERSE EVENTS:
Time Frame: Adverse events were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until LPLV (up to Day 112 (EOS))
Arm/Group | LMB763 100 mg | LMB763 50 mg | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/44 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/37 | 3/44 | 0/40
Other Adverse Events (participants affected / at risk) | 35/37 | 37/44 | 33/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LMB763 100 mg (N=37) | LMB763 50 mg (N=44) | Pooled Placebo (N=40)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LMB763 100 mg (N=37) | LMB763 50 mg (N=44) | Pooled Placebo (N=40)
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 3
Constipation (Gastrointestinal disorders) | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 3
Faeces pale (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 5 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Fatigue (General disorders) | 2 | 2 | 4
Influenza like illness (General disorders) | 4 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 4
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3
Oral herpes (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 3
Viral infection (Infections and infestations) | 0 | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 2 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 3
Blood creatinine increased (Investigations) | 3 | 1 | 0
Blood glucose increased (Investigations) | 1 | 1 | 2
Eosinophil count increased (Investigations) | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2
Lymphocyte count decreased (Investigations) | 3 | 0 | 0
Lymphocyte count increased (Investigations) | 2 | 0 | 2
Neutrophil count decreased (Investigations) | 4 | 1 | 4
Urine albumin/creatinine ratio increased (Investigations) | 2 | 4 | 5
Urine protein/creatinine ratio increased (Investigations) | 7 | 8 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 3 | 1
Headache (Nervous system disorders) | 3 | 7 | 8
Paraesthesia (Nervous system disorders) | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 2 | 0
Renal disorder (Renal and urinary disorders) | 0 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 13 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT02913105/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT02913105/SAP_001.pdf